CLINICAL TRIAL: NCT03893448
Title: A Phase 3, Multicenter, Randomized, Double-blind, Active-Comparator-controlled Study to Evaluate the Safety, Tolerability, and Immunogenicity of a 4-dose Regimen of V114 in Healthy Infants (PNEU-PED)
Brief Title: Safety, Tolerability, and Immunogenicity of V114 in Healthy Infants (V114-029)
Acronym: PNEU-PED
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V114-029; V114-029 (Other: Merck); 2018-004109-21 (EudraCT Number)
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Results first posted 2022-03-25 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Pneumococcal Infections; Pneumococcal Vaccines
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine; RotaTeq; pentacel; Recombivax HB; Hepatitis A Vaccines; Chickenpox Vaccine; Hiberix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- V114 (Experimental): Participants receive 4 total 0.5 mL intramuscular (IM) vaccinations at ~2, 4, 6, and 12 to 15 months of age. Participants will receive other vaccinations (i.e., RotaTeq™, Pentacel™, RECOMBIVAX HB™, VAQTA™, M-M-R II™, VARIVAX™, and HIBERIX™) as part of their vaccination schedule.
  Interventions: Biological: V114; Biological: RotaTeq™; Biological: Pentacel™; Biological: RECOMBIVAX HB™; Biological: VAQTA™; Biological: MMR II™; Biological: VARIVAX™; Biological: HIBERIX™
- Prevnar 13™ (Active Comparator): Participants receive 4 total 0.5 mL IM vaccinations at ~2, 4, 6, and 12 to 15 months of age. Participants will also receive other vaccines (i.e., RotaTeq™, Pentacel™, RECOMBIVAX HB™, VAQTA™, M-M-R II™, VARIVAX™, and HIBERIX™) as part of their vaccination schedule.
  Interventions: Biological: Prevnar 13™; Biological: RotaTeq™; Biological: Pentacel™; Biological: RECOMBIVAX HB™; Biological: VAQTA™; Biological: MMR II™; Biological: VARIVAX™; Biological: HIBERIX™

INTERVENTIONS:
Biological: V114 — V114 15-valent pneumococcal conjugate vaccine containing 13 serotypes present in Prevnar 13® (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) and 2 unique serotypes (22F and 33F) in each 0.5 mL intramuscular administration.
  Other Names: VAXNEUVANCE™; Pneumococcal 15-Valent Conjugate Vaccine
  Arms: V114
Biological: Prevnar 13™ — Prevnar 13™ 13-valent pneumococcal conjugate vaccine containing 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) in each 0.5 mL IM administration.
  Arms: Prevnar 13™
Biological: RotaTeq™ — A total of 3 RotaTeq™ 2 mL oral dosings at ~2, ~4, and ~6 months of age.
Biological: Pentacel™ — A total of 3 Pentacel™ 0.5 mL IM dosings at ~2, ~4, and ~6 months of age.
Biological: RECOMBIVAX HB™ — A total of 3 RECOMBIVAX HB™ 0.5 mL IM dosings at ~2, ~4, and ~6 months of age.
Biological: VAQTA™ — One VAQTA™ 0.5 mL IM dosing at 12 to 15 months of age.
Biological: MMR II™ — One MMR II™ 0.5 mL subcutaneous (SC) dosing at 12 to 15 months of age.
Biological: VARIVAX™ — One VARIVAX™ 0.5 mL SC dosing at 12 to 15 months of age.
Biological: HIBERIX™ — One HIBERIX™ 0.5 mL IM dosing at Visit 5.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and immunogenicity of V114 in healthy infants. The primary hypotheses are that: 1) V114 is non-inferior to Prevnar 13™ for the 13 shared serotypes between V114 and Prevnar 13™ based on response rates at 30 days following Dose 3; 2) V114 is non-inferior to Prevnar 13™ for the 2 unique V114 serotypes based on the response rate of the 2 unique V114 serotypes compared with the lowest response rate of any of the shared serotypes in Prevnar 13™, excluding serotype 3, at 30 days following Dose 3; 3) V114 is non-inferior to Prevnar 13™ for the 13 shared serotypes based on anti-pneumococcal polysaccharide (PnPs) serotype-specific immunoglobulin g (IgG) geometric mean concentrations (GMCs) at 30 days following Dose 3; 4) V114 is non-inferior to Prevnar 13™ for the 2 unique V114 serotypes based on the anti-PnPs serotype-specific IgG GMCs of the 2 unique V114 serotypes compared with the lowest IgG GMC of any of the shared serotypes in Prevnar 13™, excluding serotype 3, at 30 days following Dose 3; 5) V114 is non-inferior to Prevnar 13™ for the 13 shared serotypes between V114 and Prevnar 13™ based on anti-PnPs serotype-specific IgG GMCs at 30 days following Dose 4; and 6) V114 is non-inferior to Prevnar 13™ for the 2 unique V114 serotypes based on anti-PnPs serotype-specific IgG GMCs of the 2 unique V114 serotypes compared with the lowest IgG GMC of any of the shared serotypes in Prevnar 13, excluding serotype 3, at 30 days following Dose 4.

ELIGIBILITY:
Inclusion Criteria:

* Is healthy (based on a review of medical history and physical examination) in the clinical judgement of the investigator
* Has a legally acceptable representative who understands the study procedures, alternate treatments available, and risks involved with the study and voluntarily agrees to participate by giving written informed consent.

Exclusion Criteria:

* Has a history of invasive pneumococcal disease (IPD; positive blood culture, positive cerebrospinal fluid culture, or other sterile site) or known history of other culture positive pneumococcal disease.
* Has a known hypersensitivity to any component of the pneumococcal conjugate vaccine (PCV), any component of the licensed pediatric vaccines to be administered concomitantly in the study, or any diphtheria toxoid-containing vaccine.
* Has any contraindication to the concomitant study vaccines being administered in the study.
* Had a recent febrile illness (rectal temperature ≥38.1°C [=100.5°F] or axillary temperature ≥37.8°C [=100.0°F]) occurring within 72 hours prior to receipt of study vaccine.

Ages: 42 Days to 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1720 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2021-05-24 (Actual); Study Completion 2021-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (81):
- United States (66):
  - Alabama Clinical Therapeutics ( Site 0159), Birmingham, Alabama
  - Southeastern Pediatric Associates, P.A. ( Site 0107), Dothan, Alabama
  - South Alabama Pediatrics ( Site 0263), Opp, Alabama
  - Northwest Arkansas Pediatric Clinic ( Site 0172), Fayetteville, Arkansas
  - Children's Clinic of Jonesboro, PA ( Site 0184), Jonesboro, Arkansas
  - Advanced Clinical Research - Rancho Paseo ( Site 0163), Banning, California
  - Altissima Clinical Research LLC ( Site 0213), Bellflower, California
  - Southland Clinical Research Center ( Site 0187), Bellflower, California
  - Premier Health Research Center, LLC ( Site 0121), Downey, California
  - Kaiser Permanente Vaccine Study Center - Oakland ( Site 0282), Oakland, California
  - Kaiser Permanente - Sacramento ( Site 0257), Sacramento, California
  - Kaiser Permanente Vaccine Study Center - South Sacramento ( Site 0256), Sacramento, California
  - Kaiser Permanente - San Jose ( Site 0258), San Jose, California
  - Kaiser Permanente - Santa Clara ( Site 0244), Santa Clara, California
  - Davita Medical Group ( Site 0141), Colorado Springs, Colorado
  - Suncoast Research Associates, LLC ( Site 0250), Miami, Florida
  - Suncoast Research Associates, LLC ( Site 0249), North Miami Beach, Florida
  - Children's Health Center ( Site 0272), Tampa, Florida
  - Saltzer Medical Group ( Site 0215), Nampa, Idaho
  - Kentucky Pediatric/Adult Research Inc ( Site 0136), Bardstown, Kentucky
  - Michael W Simon, MD., Pediatric & Adolescent Medicine ( Site 0276), Nicholasville, Kentucky
  - ACC Pediatric Research ( Site 0147), Haughton, Louisiana
  - Medpharmics, LLC ( Site 0157), Metairie, Louisiana
  - Virgo-Carter Pediatrics ( Site 0275), Silver Spring, Maryland
  - Tufts Medical Center-Floating Hospital for Children ( Site 0129), Boston, Massachusetts
  - Pediatric Associates of Fall River ( Site 0183), Fall River, Massachusetts
  - MediSync Clinical Research Hattiesburg Clinic ( Site 0259), Petal, Mississippi
  - Children's Mercy Clinics on Broadway ( Site 0171), Kansas City, Missouri
  - Midwest Children's Health Research Institute, LLC ( Site 0109), Lincoln, Nebraska
  - Midwest Children's Health Research Institute, LLC ( Site 0106), Lincoln, Nebraska
  - Children's Physicians, UNMC ( Site 0252), Omaha, Nebraska
  - Southwest CARE Center ( Site 0161), Santa Fe, New Mexico
  - Child Health Care Associates ( Site 0242), East Syracuse, New York
  - Child Health Care Associates ( Site 0267), Liverpool, New York
  - Advantage Clinical Trials ( Site 0274), The Bronx, New York
  - Haywood Pediatric and Adolescent Medicine Group ( Site 0248), Clyde, North Carolina
  - Capitol Pediatrics & Adolescent Center ( Site 0223), Raleigh, North Carolina
  - Senders Pediatrics ( Site 0190), Cleveland, Ohio
  - Dayton Clinical Research ( Site 0188), Dayton, Ohio
  - Cyn3rgy Research ( Site 0246), Gresham, Oregon
  - Pediatric Medical Associates ( Site 0239), East Norriton, Pennsylvania
  - Allegheny Health & Wellness Pavilion West ( Site 0210), Erie, Pennsylvania
  - Lockman & Lubell Pediatrics ( Site 0166), Fort Washington, Pennsylvania
  - CCP- Kid's Way ( Site 0130), Hermitage, Pennsylvania
  - Palmetto Pediatrics, PA ( Site 0164), Charleston, South Carolina
  - Cheraw Pediatrics ( Site 0280), Cheraw, South Carolina
  - Parkside Pediatric ( Site 0125), Greenville, South Carolina
  - Holston Medical Group ( Site 0165), Kingsport, Tennessee
  - DFW Clinical Research ( Site 0111), Dallas, Texas
  - University of Texas Medical Branch ( Site 0185), Galveston, Texas
  - Ventavia Research Group LLC ( Site 0142), Houston, Texas
  - Pediatric Associates ( Site 0209), Houston, Texas
  - Houston Clinical Research Network ( Site 0266), Houston, Texas
  - Ventavia Research Group LLC ( Site 0139), Keller, Texas
  - FMC Science ( Site 0115), Lampasas, Texas
  - University of Texas Medical Branch ( Site 0170), League City, Texas
  - DCOL Center for Clinical Research ( Site 0247), Longview, Texas
  - Wee Care Pediatrics ( Site 0154), Layton, Utah
  - Cottonwood Pediatrics ( Site 0153), Murray, Utah
  - Pediatric Care ( Site 0138), Provo, Utah
  - Wee Care Pediatrics-Roy ( Site 0174), Roy, Utah
  - University of Utah ( Site 0214), Salt Lake City, Utah
  - Dixie Pediatrics ( Site 0260), St. George, Utah
  - Wee Care Pediatrics ( Site 0193), Syracuse, Utah
  - MultiCare Rockwood Cheney Clinic ( Site 0195), Cheney, Washington
  - Multicare / Rockwood Clinic ( Site 0167), Spokane, Washington
- Puerto Rico (6):
  - Cooperativa de Facultad Medica Sanacoop ( Site 0077), Bayamón
  - Clinical Research of Puerto Rico ( Site 0075), Guayama
  - CAIMED Center - Ponce School of Medicine ( Site 0076), Ponce
  - San Juan Hospital ( Site 0079), San Juan
  - University of Puerto Rico - Medical Science Campus ( Site 0078), San Juan
  - Elba Antoniette Perez Vargas MD-Private Practice ( Site 0081), Trujillo Alto
- Thailand (4):
  - Khon Kaen University ( Site 0031), Muang, Changwat Khon Kaen
  - Phramongkutklao Hospital ( Site 0033), Bangkok
  - Siriraj Hospital ( Site 0032), Bangkok
  - Maharaj Nakorn Chiang Mai Hospital ( Site 0030), Chiang Mai
- Turkey (Türkiye) (5):
  - Cukurova Uni Tip Fak Cocuk Saglıgı ve Hasta ABD ( Site 0060), Adana
  - Ankara Universitesi Tip Fakultesi ( Site 0053), Ankara
  - Ege University Medical Faculty Hospital ( Site 0050), Izmir
  - Dokuz Eylul University Faculty of Medicine ( Site 0054), Izmir
  - Erciyes Universitesi Tip Fakultesi ( Site 0057), Kayseri

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Lupinacci R, Rupp R, Wittawatmongkol O, Jones J, Quinones J, Ulukol B, Dagan R, Richmond P, Stek JE, Romero L, Koseoglu S, Tamms G, McFetridge R, Li J, Cheon K, Musey L, Banniettis N, Bickham K; V114-029 PNEU-PED study group. A phase 3, multicenter, randomized, double-blind, active-comparator-controlled study to evaluate the safety, tolerability, and immunogenicity of a 4-dose regimen of V114, a 15-valent pneumococcal conjugate vaccine, in healthy infants (PNEU-PED). Vaccine. 2023 Jan 27;41(5):1142-1152. doi: 10.1016/j.vaccine.2022.12.054. Epub 2023 Jan 6. PMID 36621410
- [Derived] Mt-Isa S, Chumbley JR, Crawford EL, Banniettis N, Buchwald UK, Weaver J, Weiss T. An indirect treatment comparison (ITC) and matching-adjusted indirect comparison (MAIC) between a 15-valent (V114) and a 20-valent (PCV20) pneumococcal conjugate vaccine among healthy infants. Expert Rev Vaccines. 2023 Jan-Dec;22(1):906-917. doi: 10.1080/14760584.2023.2270039. Epub 2023 Oct 19. PMID 37846456

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study recruited healthy infants approximately 2 months (42 to 90 days, inclusive) of age, without a history of invasive pneumococcal disease or prior administration of any pneumococcal vaccine.
Pre-assignment Details: 1720 participants were randomized in a 1:1 ratio to receive a 4-dose regimen of either V114 or Prevnar 13™. One participant randomized to the Prevnar 13™ arm was inadvertently treated with Prevnar 13™ and V114.
Groups:
- V114: Participants received a single 0.5 mL intramuscular (IM) injection of V114 on Day 1 from 42-90 days of age inclusive (Vaccination 1), Month 4 from 4 months of age to 1 day prior to 5 months of age (Vaccination 2), Month 6 from 6 months of age to 1 day prior to 7 months of age (Vaccination 3) and Months 12-15 from 12 months of age to 1 day prior to 16 months of age (Vaccination 4). Participants concomitantly received other licensed paediatric vaccines as follows: RotaTeq™, Pentacel™, RECOMBIVAX HB™ on Day 1, Month 4, and Month 6; VAQTA™, HIBERIX™, M-M-R™ II, VARIVAX™ on Months 12-15.
- Prevnar 13™: Participants received a single 0.5 mL IM injection of Prevnar 13™ on Day 1 from 42-90 days of age inclusive (Vaccination 1), Month 4 from 4 months of age to 1 day prior to 5 months of age (Vaccination 2), Month 6 from 6 months of age to 1 day prior to 7 months of age (Vaccination 3) and Months 12-15 from 12 months of age to 1 day prior to 16 months of age (Vaccination 4). Participants concomitantly received other licensed paediatric vaccines as follows: RotaTeq™, Pentacel™, RECOMBIVAX HB™ on Day 1, Month 4, and Month 6; VAQTA™, HIBERIX™, M-M-R™ II, VARIVAX™ on Months 12-15.
Period: Overall Study
Arm/Group | V114 | Prevnar 13™
Started | 860 | 860
Treated | 858 | 856
Completed | 758 | 734
Not Completed | 102 | 126
Not completed — Withdrawal by Parent/Guardian | 59 | 85
Not completed — Physician Decision | 8 | 14
Not completed — Lost to Follow-up | 34 | 27
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Prevnar 13™: Participants received a single 0.5 mL IM injection of Prevnar 13™ on Day 1 between 42-90 days of age inclusive (Vaccination 1), Month 4 from 4 months of age to 1 day prior to 5 months of age (Vaccination 2), Month 6 from 6 months of age to 1 day prior to 7 months of age (Vaccination 3) and Months 12-15 from 12 months of age to 1 day prior to 16 months of age (Vaccination 4). Participants concomitantly received other licensed paediatric vaccines as follows: RotaTeq™, Pentacel™, RECOMBIVAX HB™ on Day 1, Month 4, and Month 6; VAQTA™, HIBERIX™, M-M-R™ II, VARIVAX™ on Months 12-15.
- Total: Total of all reporting groups
Arm/Group | V114 | Prevnar 13™ | Total
Number analyzed (Participants) | 860 | 860 | 1720
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 8.4 (1.2) | 8.4 (1.3) | 8.4 (1.2)
Age, Customized [Number; unit: Participants]
  In utero | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 weeks) | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 860 | 860 | 1720
  Children (2-11 years) | 0 | 0 | 0
  Adolescents (12-17 years) | 0 | 0 | 0
  Adults (18-64 years) | 0 | 0 | 0
  From 65-84 years | 0 | 0 | 0
  85 years and over | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 397 | 428 | 825
  Male | 463 | 432 | 895
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 207 | 204 | 411
  Not Hispanic or Latino | 640 | 645 | 1285
  Unknown or Not Reported | 13 | 11 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 13 | 19
  Asian | 223 | 227 | 450
  Native Hawaiian or Other Pacific Islander | 6 | 4 | 10
  Black or African American | 52 | 53 | 105
  White | 474 | 483 | 957
  More than one race | 98 | 80 | 178
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Solicited Injection-Site Adverse Events (AEs) in V114 Versus Prevnar 13™
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited injection-site AEs consisted of swelling, redness, pain or tenderness, and hard lump.
Time Frame: Up to 14 days after each vaccination with either V114 or Prevnar 13™
Population: All randomized participants who received at least 1 dose of either V114 or Prevnar 13™. One participant in the Prevnar 13™ group inadvertently received both V114 and Prevnar 13™ and was excluded from the analysis population.
Measure: Number; unit: Percentage of participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 858 | 855
Percentage of participants
  Solicited injection site AEs | 69.0 | 69.2
  Injection site erythema (redness) | 33.7 | 38.5
  Injection site induration (hard lump) | 26.3 | 26.8
  Injection site pain (pain) | 49.8 | 46.9
  Injection site swelling (swelling) | 26.3 | 24.0
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Injection site erythema Estimated difference, CI, and p-value are calculated based on the Miettinen & Nurminen method; Test type: Other; p = 0.039, Miettinen & Nurminen; Percentage Point Difference = -4.8, 95% CI 2-sided [-9.3 to -0.2] — V114-Prevnar 13™
Statistical Analysis 2: Comparison: V114 vs Prevnar 13™; Injection site induration Estimated difference, CI, and p-value are calculated based on the Miettinen & Nurminen method; Test type: Other; p = 0.836, Miettinen & Nurminen; Percentage Point Difference = -0.4, 95% CI 2-sided [-4.6 to 3.7] — V114-Prevnar 13™
Statistical Analysis 3: Comparison: V114 vs Prevnar 13™; Injection site pain Estimated difference, CI, and p-value are calculated based on the Miettinen & Nurminen method; Test type: Other; p = 0.235, Miettinen & Nurminen; Percentage Point Difference = 2.9, 95% CI 2-sided [-1.9 to 7.6] — V114-Prevnar 13™
Statistical Analysis 4: Comparison: V114 vs Prevnar 13™; Injection site swelling Estimated difference, CI, and p-value are calculated based on the Miettinen & Nurminen method; Test type: Other; p = 0.260, Miettinen & Nurminen; Percentage Point Difference = 2.4, 95% CI 2-sided [-1.7 to 6.5] — V114-Prevnar 13™

2. Primary Outcome: Percentage of Participants With Solicited Systemic AEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited systemic AEs consisted of irritability, drowsiness, appetite lost, and hives or welts.
Time Frame: Up to 14 days after each vaccination with either V114 or Prevnar 13™
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 858 | 855
Percentage of participants
  Solicited systemic adverse events | 84.4 | 84.8
  Decreased appetite | 34.3 | 36.0
  Irritability | 76.5 | 75.4
  Somnolence (drowsiness) | 59.0 | 62.0
  Urticaria (hives) | 6.5 | 6.5
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Decreased appetite Estimated difference, CI, and p-value are calculated based on the Miettinen & Nurminen method; Test type: Other; p = 0.446, Miettinen & Nurminen; Percentage Point Difference = -1.8, 95% CI 2-sided [-6.3 to 2.8] — V114-Prevnar 13™
Statistical Analysis 2: Comparison: V114 vs Prevnar 13™; Irritability Estimated difference, CI, and p-value are calculated based on the Miettinen & Nurminen method; Test type: Other; p = 0.622, Miettinen & Nurminen; Percentage Point Difference = 1.0, 95% CI 2-sided [-3.0 to 5.1] — V114-Prevnar 13™
Statistical Analysis 3: Comparison: V114 vs Prevnar 13™; Somnolence (drowsiness) Estimated difference, CI, and p-value are calculated based on the Miettinen & Nurminen method; Test type: Other; p = 0.202, Miettinen & Nurminen; Percentage Point Difference = -3.0, 95% CI 2-sided [-7.6 to 1.6] — V114-Prevnar 13™
Statistical Analysis 4: Comparison: V114 vs Prevnar 13™; Urticaria (Hives) Estimated difference, CI, and p-value are calculated based on the Miettinen & Nurminen method; Test type: Other; p = 0.985, Miettinen & Nurminen; Percentage Point Difference = 0.0, 95% CI 2-sided [-2.4 to 2.3] — V114-Prevnar 13™

3. Primary Outcome: Percentage of Participants With Vaccine-Related Serious Adverse Events (SAEs)
Description: An SAE is any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires inpatient hospitalization or prolongs existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an other important medical event. Any SAEs that are at least possibly related to vaccination are summarized.
Time Frame: From Day 1 up to 6 months after Vaccination 4 (up to 21 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 858 | 855
Percentage of participants | 0.0 | 0.0
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Estimated difference, CI, and p-value are calculated based on the Miettinen & Nurminen method; Test type: Other; Percentage Point Difference = 0.0, 95% CI 2-sided [-0.4 to 0.4] — V114-Prevnar 13™

4. Primary Outcome: Percentage of Participants With Anti-Pneumococcal Polysaccharide (Anti-PnP) Immunoglobulin G (IgG) Antibody (Ab) ≥0.35 ug/mL One Month After Vaccination 3
Description: Anti-PnP serotype-specific IgG response rates for the 15 serotypes contained in V114 were measured with pneumococcal electrochemiluminescence (PnECL). The percentage of participants with IgG Ab ≥0.35 ug/mL are reported for each serotype.
Time Frame: One month after Vaccination 3 (Month 7)
Population: All randomized participants who did not have protocol deviations that could have substantially affected the results of the immunogenicity analysis and who had sufficient blood volume to perform the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 858 | 856
Percentage of participants
  Serotype 1: number analyzed (Participants) | 702 | 665
  Serotype 1 | 95.7 | 99.1
  Serotype 3: number analyzed (Participants) | 699 | 662
  Serotype 3 | 94.7 | 79.2
  Serotype 4: number analyzed (Participants) | 699 | 663
  Serotype 4 | 96.4 | 98.6
  Serotype 5: number analyzed (Participants) | 702 | 664
  Serotype 5 | 95.3 | 97.4
  Serotype 6A: number analyzed (Participants) | 702 | 663
  Serotype 6A | 93.7 | 98.6
  Serotype 6B: number analyzed (Participants) | 699 | 662
  Serotype 6B | 88.6 | 92.0
  Serotype 7F: number analyzed (Participants) | 701 | 665
  Serotype 7F | 99.0 | 99.8
  Serotype 9V: number analyzed (Participants) | 700 | 661
  Serotype 9V | 97.1 | 98.2
  Serotype 14: number analyzed (Participants) | 700 | 661
  Serotype 14 | 97.9 | 97.9
  Serotype 18C: number analyzed (Participants) | 700 | 662
  Serotype 18C | 97.4 | 98.3
  Serotype 19A: number analyzed (Participants) | 702 | 665
  Serotype 19A | 97.9 | 99.7
  Serotype 19F: number analyzed (Participants) | 700 | 663
  Serotype 19F | 99.0 | 100.0
  Serotype 23F: number analyzed (Participants) | 698 | 661
  Serotype 23F | 91.5 | 91.8
  Serotype 22F: number analyzed (Participants) | 701 | 661
  Serotype 22F | 98.6 | 91.8
  Serotype 33F: number analyzed (Participants) | 702 | 661
  Serotype 33F | 87.3 | 91.8
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Serotype 1 Estimated difference, CI, and p-value are calculated based on the Miettinen & Nurminen method; Test type: Non-Inferiority — A conclusion of non-inferiority of V114 to Prevnar 13™ is based on the lower bound of the 2-sided 95% CI for the difference in percentages (V114 - Prevnar 13™) being >-10 percentage points (1-sided p-value <0.025); p < 0.001, Miettinen & Nurminen — p-value is 1-sided; Percentage Point Difference = -3.4, 95% CI 2-sided [-5.2 to -1.8] — V114-Prevnar 13™
Statistical Analysis 2: Comparison: V114 vs Prevnar 13™; Serotype 3 Estimated difference, CI, and p-value are calculated based on the Miettinen & Nurminen method; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen & Nurminen — p-value is 1-sided; Percentage Point Difference = 15.6, 95% CI 2-sided [12.1 to 19.2] — V114-Prevnar 13™
Statistical Analysis 3: Comparison: V114 vs Prevnar 13™; Serotype 4 Estimated difference, CI, and p-value are calculated based on the Miettinen & Nurminen method; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen & Nurminen — p-value is 1-sided; Percentage Point Difference = -2.2, 95% CI 2-sided [-4.0 to -0.6] — V114-Prevnar 13™
Statistical Analysis 4: Comparison: V114 vs Prevnar 13™; Serotype 5 Estimated difference, CI, and p-value are calculated based on the Miettinen & Nurminen method; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen & Nurminen — p-value is 1-sided; Percentage Point Difference = -2.1, 95% CI 2-sided [-4.2 to -0.2] — V114-Prevnar 13™
Statistical Analysis 5: Comparison: V114 vs Prevnar 13™; Serotype 6A Estimated difference, CI, and p-value are calculated based on the Miettinen & Nurminen method; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen & Nurminen — p-value is 1-sided; Percentage Point Difference = -4.9, 95% CI 2-sided [-7.1 to -3.0] — V114-Prevnar 13™
Statistical Analysis 6: Comparison: V114 vs Prevnar 13™; Serotype 6B Estimated difference, CI, and p-value are calculated based on the Miettinen & Nurminen method; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen & Nurminen — p-value is 1-sided; Percentage Point Difference = -3.4, 95% CI 2-sided [-6.6 to -0.3] — V114-Prevnar 13™
Statistical Analysis 7: Comparison: V114 vs Prevnar 13™; Serotype 7F Estimated difference, CI, and p-value are calculated based on the Miettinen & Nurminen method; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen & Nurminen — p-value is 1-sided; Percentage Point Difference = -0.8, 95% CI 2-sided [-1.9 to -0.1] — V114-Prevnar 13™
Statistical Analysis 8: Comparison: V114 vs Prevnar 13™; Serotype 9V Estimated difference, CI, and p-value are calculated based on the Miettinen & Nurminen method; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen & Nurminen — p-value is 1-sided; Percentage Point Difference = -1.0, 95% CI 2-sided [-2.8 to 0.6] — V114-Prevnar 13™
Statistical Analysis 9: Comparison: V114 vs Prevnar 13™; Serotype 14 Estimated difference, CI, and p-value are calculated based on the Miettinen & Nurminen method; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen & Nurminen — p-value is 1-sided; Percentage Point Difference = 0.0, 95% CI 2-sided [-1.6 to 1.6] — V114-Prevnar 13™
Statistical Analysis 10: Comparison: V114 vs Prevnar 13™; Serotype 18C Estimated difference, CI, and p-value are calculated based on the Miettinen & Nurminen method; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen & Nurminen — p-value is 1-sided; Percentage Point Difference = -0.9, 95% CI 2-sided [-2.6 to 0.7] — V114-Prevnar 13™
Statistical Analysis 11: Comparison: V114 vs Prevnar 13™; Serotype 19A Estimated difference, CI, and p-value are calculated based on the Miettinen & Nurminen method; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen & Nurminen — p-value is 1-sided; Percentage Point Difference = -1.8, 95% CI 2-sided [-3.2 to -0.8] — V114-Prevnar 13™
Statistical Analysis 12: Comparison: V114 vs Prevnar 13™; Serotype 19F Estimated difference, CI, and p-value are calculated based on the Miettinen & Nurminen method; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen & Nurminen — p-value is 1-sided; Percentage Point Difference = -1.0, 95% CI 2-sided [-2.1 to -0.4] — V114-Prevnar 13™
Statistical Analysis 13: Comparison: V114 vs Prevnar 13™; Serotype 23F Estimated difference, CI, and p-value are calculated based on the Miettinen & Nurminen method; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen & Nurminen — p-value is 1-sided; Percentage Point Difference = -0.3, 95% CI 2-sided [-3.2 to 2.7] — V114-Prevnar 13™
Statistical Analysis 14: Comparison: V114 vs Prevnar 13™; Serotype 22F This analysis represents the difference between response rate to Serotype 22F in recipients of V114 and lowest response (Serotype 23F at 91.8) in recipients of Prevnar 13™ for shared serotypes, excluding serotype 3. Estimated difference, CI, and p-value are calculated based on the Miettinen & Nurminen method; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen & Nurminen — p-value is 1-sided; Percentage Point Difference = 6.7, 95% CI 2-sided [4.6 to 9.2] — V114-Prevnar 13™
Statistical Analysis 15: Comparison: V114 vs Prevnar 13™; Serotype 33F This analysis represents the difference between response rate to Serotype 33F in recipients of V114 and lowest response (Serotype 23F at 91.8) in recipients of Prevnar 13™ for shared serotypes, excluding serotype 3. Estimated difference, CI, and p-value are calculated based on the Miettinen & Nurminen method; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen & Nurminen — p-value is 1-sided; Percentage Point Difference = -4.5, 95% CI 2-sided [-7.8 to -1.3] — V114-Prevnar 13™

5. Primary Outcome: Geometric Mean Concentration (GMC) of Anti-PnP IgG Ab One Month After Vaccination 3
Description: The GMC of anti-PnP IgG Ab were measured with PnECL one month after vaccination 3 and reported for the 15 serotypes contained in V114. IgG GMCs were compared to the lowest in recipients of Prevnar 13™ excluding serotype 3 for the 2 serotypes unique to V114, and compared to the same serotypes for the 13 shared serotypes.
Time Frame: One month after Vaccination 3 (Month 7)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 858 | 856
ug/mL
  Serotype 1: number analyzed (Participants) | 702 | 665
  Serotype 1 | 1.21 [1.15 to 1.27] | 1.89 [1.79 to 2.00]
  Serotype 3: number analyzed (Participants) | 699 | 662
  Serotype 3 | 1.08 [1.03 to 1.14] | 0.62 [0.59 to 0.66]
  Serotype 4: number analyzed (Participants) | 699 | 663
  Serotype 4 | 1.29 [1.22 to 1.36] | 1.35 [1.28 to 1.43]
  Serotype 5: number analyzed (Participants) | 702 | 664
  Serotype 5 | 1.63 [1.52 to 1.74] | 2.25 [2.09 to 2.41]
  Serotype 6A: number analyzed (Participants) | 702 | 663
  Serotype 6A | 1.55 [1.44 to 1.66] | 2.95 [2.76 to 3.15]
  Serotype 6B: number analyzed (Participants) | 699 | 662
  Serotype 6B | 1.60 [1.45 to 1.76] | 1.97 [1.80 to 2.16]
  Serotype 7F: number analyzed (Participants) | 701 | 665
  Serotype 7F | 2.48 [2.35 to 2.61] | 3.23 [3.06 to 3.40]
  Serotype 9V: number analyzed (Participants) | 700 | 661
  Serotype 9V | 1.73 [1.63 to 1.83] | 1.89 [1.77 to 2.01]
  Serotype 14: number analyzed (Participants) | 700 | 661
  Serotype 14 | 4.78 [4.44 to 5.16] | 6.80 [6.30 to 7.33]
  Serotype 18C: number analyzed (Participants) | 700 | 662
  Serotype 18C | 1.53 [1.44 to 1.61] | 2.00 [1.88 to 2.13]
  Serotype 19A: number analyzed (Participants) | 702 | 665
  Serotype 19A | 1.63 [1.54 to 1.73] | 2.29 [2.16 to 2.44]
  Serotype 19F: number analyzed (Participants) | 700 | 663
  Serotype 19F | 2.01 [1.91 to 2.11] | 2.72 [2.59 to 2.86]
  Serotype 23F: number analyzed (Participants) | 698 | 661
  Serotype 23F | 1.31 [1.22 to 1.41] | 1.47 [1.36 to 1.59]
  Serotype 22F: number analyzed (Participants) | 701 | 660
  Serotype 22F | 4.91 [4.58 to 5.26] | 0.05 [0.05 to 0.06]
  Serotype 33F: number analyzed (Participants) | 702 | 664
  Serotype 33F | 1.67 [1.51 to 1.85] | 0.06 [0.05 to 0.06]
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Serotype 1 GMC ratio, CI, and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — A conclusion of non-inferiority of V114 to Prevnar 13™ is based on the lower bound of the 2-sided 95% CI for the GMC ratio (V114/Prevnar 13™) being >0.5 (1-sided p-value <0.025); p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 0.64, 95% CI 2-sided [0.59 to 0.69] — V114/Prevnar 13™
Statistical Analysis 2: Comparison: V114 vs Prevnar 13™; Serotype 3 GMC ratio, CI, and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 1.73, 95% CI 2-sided [1.61 to 1.87] — V114/Prevnar 13™
Statistical Analysis 3: Comparison: V114 vs Prevnar 13™; Serotype 4 GMC ratio, CI, and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 0.95, 95% CI 2-sided [0.88 to 1.03] — V114/Prevnar 13™
Statistical Analysis 4: Comparison: V114 vs Prevnar 13™; Serotype 5 GMC ratio, CI, and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 0.72, 95% CI 2-sided [0.66 to 0.80] — V114/Prevnar 13™
Statistical Analysis 5: Comparison: V114 vs Prevnar 13™; Serotype 6A GMC ratio, CI, and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p = 0.167, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 0.52, 95% CI 2-sided [0.48 to 0.58] — V114/Prevnar 13™
Statistical Analysis 6: Comparison: V114 vs Prevnar 13™; Serotype 6B GMC ratio, CI, and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 0.81, 95% CI 2-sided [0.71 to 0.93] — V114/Prevnar 13™
Statistical Analysis 7: Comparison: V114 vs Prevnar 13™; Serotype 7F GMC ratio, CI, and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 0.77, 95% CI 2-sided [0.71 to 0.83] — V114/Prevnar 13™
Statistical Analysis 8: Comparison: V114 vs Prevnar 13™; Serotype 9V GMC ratio, CI, and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 0.91, 95% CI 2-sided [0.84 to 1.00] — V114/Prevnar 13™
Statistical Analysis 9: Comparison: V114 vs Prevnar 13™; Serotype 14 GMC ratio, CI, and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 0.70, 95% CI 2-sided [0.63 to 0.78] — V114/Prevnar 13™
Statistical Analysis 10: Comparison: V114 vs Prevnar 13™; Serotype 18C GMC ratio, CI, and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 0.76, 95% CI 2-sided [0.70 to 0.83] — V114/Prevnar 13™
Statistical Analysis 11: Comparison: V114 vs Prevnar 13™; Serotype 19A GMC ratio, CI, and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 0.71, 95% CI 2-sided [0.65 to 0.77] — V114/Prevnar 13™
Statistical Analysis 12: Comparison: V114 vs Prevnar 13™; Serotype 19F GMC ratio, CI, and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 0.74, 95% CI 2-sided [0.69 to 0.79] — V114/Prevnar 13™
Statistical Analysis 13: Comparison: V114 vs Prevnar 13™; Serotype 23F GMC ratio, CI, and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 0.89, 95% CI 2-sided [0.80 to 0.99] — V114/Prevnar 13™
Statistical Analysis 14: Comparison: V114 vs Prevnar 13™; Serotype 22F IgG GMC for Serotype 22F in recipients of V114 was compared to lowest IgG GMC (Serotype 4 at 1.35 ug/mL) for shared serotype in recipients of Prevnar 13™, excluding serotype 3. GMC ratio, CI, and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 3.64, 95% CI 2-sided [3.33 to 3.98] — V114/Prevnar 13™
Statistical Analysis 15: Comparison: V114 vs Prevnar 13™; Serotype 33F IgG GMC for Serotype 33F in recipients of V114 was compared to lowest IgG GMC (Serotype 4 at 1.35 ug/mL) for shared serotype in recipients of Prevnar 13™, excluding serotype 3. GMC ratio, CI, and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 1.24, 95% CI 2-sided [1.10 to 1.39] — V114/Prevnar 13™

6. Primary Outcome: GMC of Anti-PnP IgG Ab One Month After Vaccination 4
Description: The GMC of anti-PnP IgG Ab were measured with PnECL one month after vaccination 4 and reported for the 15 serotypes contained in V114. IgG GMCs were compared to the lowest in recipients of Prevnar 13™ excluding serotype 3 for the 2 serotypes unique to V114, and compared to the same serotypes for the 13 shared serotypes.
Time Frame: One month after Vaccination 4 (Month 13 to Month 16)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 858 | 856
ug/mL
  Serotype 1: number analyzed (Participants) | 715 | 685
  Serotype 1 | 1.35 [1.27 to 1.42] | 2.03 [1.92 to 2.14]
  Serotype 3: number analyzed (Participants) | 712 | 686
  Serotype 3 | 0.96 [0.91 to 1.01] | 0.71 [0.67 to 0.75]
  Serotype 4: number analyzed (Participants) | 713 | 682
  Serotype 4 | 1.23 [1.16 to 1.31] | 1.60 [1.51 to 1.71]
  Serotype 5: number analyzed (Participants) | 713 | 682
  Serotype 5 | 2.49 [2.34 to 2.64] | 3.95 [3.71 to 4.20]
  Serotype 6A: number analyzed (Participants) | 713 | 682
  Serotype 6A | 3.70 [3.46 to 3.97] | 6.21 [5.83 to 6.62]
  Serotype 6B: number analyzed (Participants) | 712 | 682
  Serotype 6B | 4.76 [4.43 to 5.10] | 6.43 [6.02 to 6.88]
  Serotype 7F: number analyzed (Participants) | 714 | 686
  Serotype 7F | 3.42 [3.22 to 3.64] | 4.85 [4.56 to 5.16]
  Serotype 9V: number analyzed (Participants) | 716 | 686
  Serotype 9V | 2.40 [2.27 to 2.55] | 3.29 [3.10 to 3.49]
  Serotype 14: number analyzed (Participants) | 716 | 685
  Serotype 14 | 5.61 [5.21 to 6.04] | 6.95 [6.51 to 7.43]
  Serotype 18C: number analyzed (Participants) | 713 | 684
  Serotype 18C | 2.62 [2.46 to 2.78] | 3.08 [2.88 to 3.29]
  Serotype 19A: number analyzed (Participants) | 715 | 685
  Serotype 19A | 4.10 [3.88 to 4.33] | 5.53 [5.21 to 5.87]
  Serotype 19F: number analyzed (Participants) | 715 | 685
  Serotype 19F | 3.55 [3.37 to 3.75] | 4.47 [4.23 to 4.73]
  Serotype 23F: number analyzed (Participants) | 713 | 683
  Serotype 23F | 2.04 [1.91 to 2.18] | 3.32 [3.08 to 3.58]
  Serotype 22F: number analyzed (Participants) | 714 | 682
  Serotype 22F | 7.52 [7.09 to 7.98] | 0.11 [0.10 to 0.12]
  Serotype 33F: number analyzed (Participants) | 714 | 677
  Serotype 33F | 4.15 [3.89 to 4.42] | 0.09 [0.09 to 0.10]
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Serotype 1 GMC ratio, CI, and p-value are calculated using the t-distribution with the variance estimate from a serotype specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 0.66, 95% CI 2-sided [0.62 to 0.72] — V114/Prevnar 13™
Statistical Analysis 2: Comparison: V114 vs Prevnar 13™; [analysis description as in outcome 5, analysis 2]; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 1.35, 95% CI 2-sided [1.25 to 1.46] — V114/Prevnar 13™
Statistical Analysis 3: Comparison: V114 vs Prevnar 13™; [analysis description as in outcome 5, analysis 3]; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 0.77, 95% CI 2-sided [0.71 to 0.84] — V114/Prevnar 13™
Statistical Analysis 4: Comparison: V114 vs Prevnar 13™; [analysis description as in outcome 5, analysis 4]; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 0.63, 95% CI 2-sided [0.58 to 0.69] — V114/Prevnar 13™
Statistical Analysis 5: Comparison: V114 vs Prevnar 13™; [analysis description as in outcome 5, analysis 5]; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 0.60, 95% CI 2-sided [0.54 to 0.65] — V114/Prevnar 13™
Statistical Analysis 6: Comparison: V114 vs Prevnar 13™; [analysis description as in outcome 5, analysis 6]; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 0.74, 95% CI 2-sided [0.67 to 0.81] — V114/Prevnar 13™
Statistical Analysis 7: Comparison: V114 vs Prevnar 13™; [analysis description as in outcome 5, analysis 7]; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 0.70, 95% CI 2-sided [0.65 to 0.77] — V114/Prevnar 13™
Statistical Analysis 8: Comparison: V114 vs Prevnar 13™; [analysis description as in outcome 5, analysis 8]; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 0.73, 95% CI 2-sided [0.67 to 0.80] — V114/Prevnar 13™
Statistical Analysis 9: Comparison: V114 vs Prevnar 13™; [analysis description as in outcome 5, analysis 9]; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 0.81, 95% CI 2-sided [0.73 to 0.89] — V114/Prevnar 13™
Statistical Analysis 10: Comparison: V114 vs Prevnar 13™; [analysis description as in outcome 5, analysis 10]; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 0.85, 95% CI 2-sided [0.78 to 0.93] — V114/Prevnar 13™
Statistical Analysis 11: Comparison: V114 vs Prevnar 13™; [analysis description as in outcome 5, analysis 11]; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 0.74, 95% CI 2-sided [0.68 to 0.80] — V114/Prevnar 13™
Statistical Analysis 12: Comparison: V114 vs Prevnar 13™; [analysis description as in outcome 5, analysis 12]; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 0.79, 95% CI 2-sided [0.74 to 0.86] — V114/Prevnar 13™
Statistical Analysis 13: Comparison: V114 vs Prevnar 13™; [analysis description as in outcome 5, analysis 13]; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 0.61, 95% CI 2-sided [0.56 to 0.68] — V114/Prevnar 13™
Statistical Analysis 14: Comparison: V114 vs Prevnar 13™; Serotype 22F IgG GMC for Serotype 22F in recipients of V114 was compared to the lowest IgG GMC (Serotype 4 at 1.60 ug/mL) for shared serotype in recipients of Prevnar 13™, excluding serotype 3. GMC ratio, CI, and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 4.69, 95% CI 2-sided [4.30 to 5.11] — V114/Prevnar 13™
Statistical Analysis 15: Comparison: V114 vs Prevnar 13™; Serotype 33F IgG GMC for Serotype 33F in recipients of V114 was compared to the lowest IgG GMC (Serotype 4 at 1.60 ug/mL) for shared serotype in recipients of Prevnar 13™, excluding serotype 3. GMC ratio, CI, and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 2.59, 95% CI 2-sided [2.36 to 2.83] — V114/Prevnar 13™

7. Secondary Outcome: Percentage of Participants Meeting Response Rate Criteria for Pentacel™-Specific (Anti-Diptheria Toxoid, Tetanus Toxoid, and Pertussis Antigens) Immunoglobulin G (IgG) Antibody (Ab) Geometric Mean Concentration (GMC) One Month After Vaccination 3
Description: Antibody responses to diphtheria toxoid, tetanus toxoid, and pertussis antigens were measured using Luminex Assay. The percentage of participants meeting specific criteria are summarized for each serotype. The serotype-specific response rate criteria are as follows: diphtheria toxoid: % ≥0.1 IU/mL; tetanus toxoid: % ≥0.1 IU/mL; pertussis toxin (PT): % ≥ 5 EU/mL; pertussis filamentous hemagglutinin (FHA): % ≥5 EU/mL; pertussis fimbrae types 2/3 (FIM 2/3): % ≥20 EU/mL; pertussis pertactin (PRN): % ≥5 EU/mL; poliovirus 1: % neutralizing antibody (NAb) ≥1:8 dilution; poliovirus 2: % NAb ≥1:8 dilution, poliovirus 3: % NAb ≥1:8 dilution; and Haemophilus influenzae Type B polyribosylribitol phosphate (Hib-PRP): % ≥0.15 ug/mL.
Time Frame: One month after Vaccination 3 (Month 7)
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 858 | 856
Percentage of participants
  Diphtheria toxoid: number analyzed (Participants) | 703 | 666
  Diphtheria toxoid | 96.9 | 97.6
  Tetanus toxoid: number analyzed (Participants) | 703 | 666
  Tetanus toxoid | 100.0 | 99.8
  Pertussis toxin: number analyzed (Participants) | 703 | 666
  Pertussis toxin | 99.0 | 98.5
  Pertussis filamentous hemagglutinin: number analyzed (Participants) | 703 | 666
  Pertussis filamentous hemagglutinin | 99.1 | 99.4
  Pertussis fimbrae types 2/3: number analyzed (Participants) | 703 | 666
  Pertussis fimbrae types 2/3 | 63.7 | 61.7
  Pertussis pertactin: number analyzed (Participants) | 703 | 666
  Pertussis pertactin | 67.3 | 65.5
  Poliovirus 1: number analyzed (Participants) | 662 | 619
  Poliovirus 1 | 99.8 | 99.8
  Poliovirus 2: number analyzed (Participants) | 648 | 614
  Poliovirus 2 | 100.0 | 100.0
  Poliovirus 3: number analyzed (Participants) | 650 | 607
  Poliovirus 3 | 100.0 | 100.0
  Hib-PRP: number analyzed (Participants) | 648 | 615
  Hib-PRP | 92.1 | 93.5
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Diphtheria toxoid % ≥0.1 IU/mL Estimated difference, CI, and p-value are based on the Miettinen & Nurminen method; Test type: Non-Inferiority — A conclusion of non-inferiority of Pentacel™ administered concomitantly with V114 to Pentacel™ administered concomitantly with Prevnar 13™ is based on the lower bound of the 2-sided 95% CI for the difference in percentages (V114 - Prevnar 13™) being greater than -10% (1-sided p-value <0.025); p < 0.001, Miettinen & Nurminen — p-value is 1-sided; Percentage Point Difference = -0.7, 95% CI 2-sided [-2.6 to 1.1] — V114-Prevnar 13™
Statistical Analysis 2: Comparison: V114 vs Prevnar 13™; Tetanus toxoid: % ≥0.1 IU/mL Estimated difference, CI, and p-value are based on the Miettinen & Nurminen method; Test type: Non-Inferiority — A conclusion of non-inferiority of Pentacel™ administered concomitantly with V114 to Pentacel™ administered concomitantly with Prevnar 13™ is based on the lower bound of the 2-sided 95% CI for the difference in percentages (V114 - Prevnar 13™) being greater than -5% (1-sided p-value <0.025); p < 0.001, Miettinen & Nurminen — p-value is 1-sided; Percentage Point Difference = 0.2, 95% CI 2-sided [-0.4 to 0.8] — V114-Prevnar 13™
Statistical Analysis 3: Comparison: V114 vs Prevnar 13™; Pertussis toxin (PT): % ≥ 5 EU/mL Estimated difference, CI, and p-value are based on the Miettinen & Nurminen method; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; p < 0.001, Miettinen & Nurminen — p-value is 1-sided; Percentage Point Difference = 0.5, 95% CI 2-sided [-0.7 to 1.9] — V114-Prevnar 13™
Statistical Analysis 4: Comparison: V114 vs Prevnar 13™; Pertussis filamentous hemagglutinin (FHA): % ≥5 EU/mL Estimated difference, CI, and p-value are based on the Miettinen & Nurminen method; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; p < 0.001, Miettinen & Nurminen — p-value is 1-sided; Percentage Point Difference = -0.3, 95% CI 2-sided [-1.3 to 0.8] — V114-Prevnar 13™
Statistical Analysis 5: Comparison: V114 vs Prevnar 13™; Pertussis fimbrae types 2/3 (FIM 2/3): % ≥20 EU/mL Estimated difference, CI, and p-value are based on the Miettinen & Nurminen method; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; p < 0.001, Miettinen & Nurminen — p-value is 1-sided; Percentage Point Difference = 2.0, 95% CI 2-sided [-3.1 to 7.1] — V114-Prevnar 13™
Statistical Analysis 6: Comparison: V114 vs Prevnar 13™; Pertussis pertactin (PRN): % ≥5 EU/mL Estimated difference, CI, and p-value are based on the Miettinen & Nurminen method; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; p < 0.001, Miettinen & Nurminen — p-value is 1-sided; Percentage Point Difference = 1.8, 95% CI 2-sided [-3.2 to 6.8] — V114-Prevnar 13™
Statistical Analysis 7: Comparison: V114 vs Prevnar 13™; Poliovirus 1: % NAb ≥1:8 dilution Estimated difference, CI, and p-value are based on the Miettinen & Nurminen method; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 2]; p < 0.001, Miettinen & Nurminen — p-value is 1-sided; Percentage Point Difference = 0.0, 95% CI 2-sided [-0.7 to 0.8] — V114-Prevnar 13™
Statistical Analysis 8: Comparison: V114 vs Prevnar 13™; Poliovirus 2: % NAb ≥1:8 dilution Estimated difference, CI, and p-value are based on the Miettinen & Nurminen method; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 2]; p < 0.001, Miettinen & Nurminen — p-value is 1-sided; Percentage Point Difference = 0.0, 95% CI 2-sided [-0.6 to 0.6] — V114-Prevnar 13™
Statistical Analysis 9: Comparison: V114 vs Prevnar 13™; Poliovirus 3: % NAb ≥1:8 dilution Estimated difference, CI, and p-value are based on the Miettinen & Nurminen method; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 2]; p < 0.001, Miettinen & Nurminen — p-value is 1-sided; Percentage Point Difference = 0.0, 95% CI 2-sided [-0.6 to 0.6] — V114-Prevnar 13™
Statistical Analysis 10: Comparison: V114 vs Prevnar 13™; Haemophilus influenzae Type B polyribosylribitol phosphate (Hib-PRP): % ≥0.15 ug/mL Estimated difference, CI, and p-value are based on the Miettinen & Nurminen method; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; p < 0.001, Miettinen & Nurminen — p-value is 1-sided; Percentage Point Difference = -1.4, 95% CI 2-sided [-4.3 to 1.5] — V114-Prevnar 13™

8. Secondary Outcome: Pertussis Antigen Immunoglobulin G (IgG) Antibody (Ab) Geometric Mean Concentration (GMC) One Month After Vaccination 3
Description: Pertussis antibody GMCs were measured using Luminex Assay.
Time Frame: One month after Vaccination 3 (Month 7)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 858 | 856
ug/mL
  Pertussis - PT: number analyzed (Participants) | 703 | 666
  Pertussis - PT | 43.73 [NA to NA] — Within-group confidence intervals (CIs) were not calculated, per protocol. | 44.35 [NA to NA] — Within-group CIs were not calculated, per protocol.
  Pertussis - FHA: number analyzed (Participants) | 703 | 666
  Pertussis - FHA | 67.51 [NA to NA] — Within-group CIs were not calculated, per protocol. | 69.18 [NA to NA] — Within-group CIs were not calculated, per protocol.
  Pertussis - FIM 2/3: number analyzed (Participants) | 703 | 666
  Pertussis - FIM 2/3 | 39.79 [NA to NA] — Within-group CIs were not calculated, per protocol. | 36.87 [NA to NA] — Within-group CIs were not calculated, per protocol.
  Pertussis - PRN: number analyzed (Participants) | 703 | 666
  Pertussis - PRN | 13.16 [NA to NA] — Within-group CIs were not calculated, per protocol. | 13.17 [NA to NA] — Within-group CIs were not calculated, per protocol.
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Pertussis - PT GMC ratio, CI, and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — A conclusion of non-inferiority of Pentacel™ administered concomitantly with V114 to Pentacel™ administered concomitantly with Prevnar 13™ is based on the lower bound of the 2-sided 95% CI for the GMC ratio (V114/Prevnar 13™) being >0.67 (1-sided p-value <0.025); p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 0.99, 95% CI 2-sided [0.89 to 1.09] — V114/Prevnar 13™
Statistical Analysis 2: Comparison: V114 vs Prevnar 13™; Pertussis - FHA GMC ratio, CI, and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — [test comment as in outcome 8, analysis 1]; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 0.98, 95% CI 2-sided [0.87 to 1.09] — V114/Prevnar 13™
Statistical Analysis 3: Comparison: V114 vs Prevnar 13™; Pertussis - FIM 2/3 GMC ratio, CI, and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — [test comment as in outcome 8, analysis 1]; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 1.08, 95% CI 2-sided [0.91 to 1.28] — V114/Prevnar 13™
Statistical Analysis 4: Comparison: V114 vs Prevnar 13™; Pertussis - PRN GMC ratio, CI, and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Non-Inferiority — [test comment as in outcome 8, analysis 1]; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 1.00, 95% CI 2-sided [0.84 to 1.19] — V114/Prevnar 13™

9. Secondary Outcome: Hepatitis A Antibody Response Rate One Month After Vaccination 4
Description: Antibody response rates to hepatitis A were measured with hepatitis A virus enzyme immunoassay (HAV EIA). The percentage of participants with hepatitis A antigen ≥10 mIU/mL are reported.
Time Frame: One month after Vaccination 4 (Month 13 to Month 16)
Population: All randomized participants who did not have protocol deviations that could have substantially affected the results of the immunogenicity analysis, who had sufficient blood volume to perform the analysis, and who had available HAV EIA data.
Measure: Number; unit: Percentage of participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 649 | 626
Percentage of participants | 97.4 | 97.1
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Estimated difference, CI, and p-value are based on the Miettinen & Nurminen method; Test type: Non-Inferiority — A conclusion of non-inferiority of VAQTA™ administered concomitantly with V114 to VAQTA™ administered concomitantly with Prevnar 13™ is based on the lower bound of the 2-sided 95% CI for the difference in percentages (V114 - Prevnar 13™) being greater than -10% (1-sided p-value <0.025); p < 0.001, Miettinen & Nurminen — p value is 1-sided; Percentage Point Difference = 0.3, 95% CI 2-sided [-1.6 to 2.2] — V114-Prevnar 13™

10. Secondary Outcome: Measles, Mumps, and Rubella Antibody Response Rate One Month After Vaccination 4
Description: Antibody responses to measles were measured with the bulk measles IgG enzyme immunoassay (EIA). Antibody responses to mumps were measured with enzyme-linked immunosorbent assay (ELISA). Antibody responses to rubella were measured with Bulk Rubella IgG EIA. The percentage of participants with measles antigen ≥255 mIU/ML; mumps antigen ≥10 mumps Ab units/mL; and rubella antigen ≥10 IU/mL, are reported.
Time Frame: One month after Vaccination 4 (Month 13 to Month 16)
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 858 | 856
Percentage of participants
  Measles antigen ≥255 mIU/ML: number analyzed (Participants) | 670 | 648
  Measles antigen ≥255 mIU/ML | 98.1 | 98.3
  Mumps antigen ≥10 mumps Ab units/mL: number analyzed (Participants) | 670 | 648
  Mumps antigen ≥10 mumps Ab units/mL | 95.8 | 97.5
  Rubella antigen ≥10 IU/mL: number analyzed (Participants) | 670 | 648
  Rubella antigen ≥10 IU/mL | 98.1 | 98.9
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Measles antigen ≥255 mIU/mL Estimated difference, CI, and p-value are based on the Miettinen & Nurminen method; Test type: Non-Inferiority — A conclusion of non-inferiority of M-M-R™ II administered concomitantly with V114 to M-M-R™ II administered concomitantly with Prevnar 13™ is based on the lower bound of the 2-sided 95% CI for the difference in percentages (V114 - Prevnar 13™) being greater than -5% (1-sided p-value <0.025); p < 0.001, Miettinen & Nurminen — p-value is 1-sided; Percentage Point Difference = -0.2, 95% CI 2-sided [-1.8 to 1.3] — V114-Prevnar 13™
Statistical Analysis 2: Comparison: V114 vs Prevnar 13™; Mumps antigen ≥10 mumps Ab units/mL Estimated difference, CI, and p-value are based on the Miettinen & Nurminen method; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; p < 0.001, Miettinen & Nurminen — p-value is 1-sided; Percentage Point Difference = -1.7, 95% CI 2-sided [-3.8 to 0.2] — V114-Prevnar 13™
Statistical Analysis 3: Comparison: V114 vs Prevnar 13™; Rubella antigen ≥10 IU/mL Estimated difference, CI, and p-value are based on the Miettinen & Nurminen method; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; p < 0.001, Miettinen & Nurminen — p-value is 1-sided; Percentage Point Difference = -0.9, 95% CI 2-sided [-2.3 to 0.5] — V114-Prevnar 13™

11. Secondary Outcome: Varicella-Zoster Virus (VZV) Antibody Response Rate One Month After Vaccination 4
Description: Antibody responses to varicella-zoster virus were measured with glycoprotein enzyme-linked immunosorbent assay (gpELISA). The percentage of participants with VZV antigen ≥5 gpELISA units/mL are reported.
Time Frame: One month after Vaccination 4 (Month 13 to Month 16)
Population: All randomized participants who did not have protocol deviations that could have substantially affected the results of the immunogenicity analysis, who had sufficient blood volume to perform the analysis, and who had available VZV gpELISA data.
Measure: Number; unit: Percentage of participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 715 | 685
Percentage of participants | 96.4 | 97.7
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Estimated difference, CI, and p-value are based on the Miettinen & Nurminen method; Test type: Non-Inferiority — A conclusion of non-inferiority of VARIVAX™ administered concomitantly with V114 to VARIVAX™ administered concomitantly with Prevnar 13™ is based on the lower bound of the 2-sided 95% CI for the difference in percentages (V114 - Prevnar 13™) being greater than -10% (1-sided p-value <0.025); p < 0.001, Miettinen & Nurminen — p-value is 1-sided; Percentage Point Difference = -1.3, 95% CI 2-sided [-3.2 to 0.5] — V114-Prevnar 13™

12. Secondary Outcome: Haemophilus Influenzae Type B Antibody Response Rate One Month After Vaccination 4
Description: Antibody responses to Haemophilus influenzae Type B polyribosylribitol phosphate (Hib PRP) were measured with ELISA. The percentage of participants with anti-HiB PRP antigen ≥0.15 ug/mL are reported.
Time Frame: One month after Vaccination 4 (Month 13 to Month 16)
Population: All randomized participants who did not have protocol deviations that could have substantially affected the results of the immunogenicity, who had sufficient blood volume to perform the analysis, and who had available Hib PRP ELISA data.
Measure: Number; unit: Percentage of participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 650 | 626
Percentage of participants | 98.9 | 100.0
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Estimated difference, CI, and p-value are based on the Miettinen & Nurminen method; Test type: Non-Inferiority — A conclusion of non-inferiority of HIBERIX™ administered concomitantly with V114 to HIBERIX™ administered concomitantly with Prevnar 13™ is based on the lower bound of the 2-sided 95% CI for the difference in percentages (V114 - Prevnar 13™) being greater than -10% (1-sided p-value <0.025); p < 0.001, Miettinen & Nurminen — p-value is 1-sided; Percentage Point Difference = -1.1, 95% CI 2-sided [-2.2 to -0.5] — V114-Prevnar 13™

13. Secondary Outcome: Anti-Pneumococcal Polysaccharide (Anti-PnP) Serotype-Specific Immunoglobulin G (IgG) Geometric Mean Concentration (GMC) One Month After Vaccination 3 for 2 Unique V114 Seroptypes
Description: Serotype-specific anti-PnP IgG GMCs for the 2 unique V114 serotypes were measured with PnECL. The GMCs for each serotype are reported.
Time Frame: One month after Vaccination 3 (Month 7)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 858 | 856
ug/mL
  22F: number analyzed (Participants) | 701 | 660
  22F | 4.91 [4.58 to 5.26] | 0.05 [0.05 to 0.06]
  33F: number analyzed (Participants) | 702 | 664
  33F | 1.67 [1.51 to 1.85] | 0.06 [0.05 to 0.06]
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Serotype 22F GMC ratio, CI, and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Superiority; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 92.03, 95% CI 2-sided [83.47 to 101.47] — V114/Prevnar 13™
Statistical Analysis 2: Comparison: V114 vs Prevnar 13™; Serotype 33F GMC ratio, CI, and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Superiority; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 29.50, 95% CI 2-sided [26.16 to 33.26] — V114/Prevnar 13™

14. Secondary Outcome: Anti-Pneumococcal Polysaccharide (Anti-PnP) Serotype-Specific Immunoglobulin G (IgG) Response Rates One Month After Vaccination 3 for 2 Unique V114 Seroptypes
Description: Serotype-specific anti-PnP IgG response rates for the 2 unique V114 serotypes were measured with PnECL. The percentage of participants with IgG Ab ≥0.35 ug/mL are reported for each serotype.
Time Frame: One month after Vaccination 3 (Month 7)
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 858 | 856
Percentage of participants
  Serotype 22F: number analyzed (Participants) | 701 | 660
  Serotype 22F | 98.6 | 3.5
  Serotype 33F: number analyzed (Participants) | 702 | 664
  Serotype 33F | 87.3 | 2.1
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Serotype 22F Estimated difference, CI, and p-value are based on the Miettinen & Nurminen method; Test type: Superiority; p < 0.001, Miettinen & Nurminen — p-value is 1-sided; Percentage Point Difference = 95.1, 95% CI 2-sided [93.1 to 96.5] — V114-Prevnar 13™
Statistical Analysis 2: Comparison: V114 vs Prevnar 13™; Serotype 33F Estimated difference, CI, and p-value are based on the Miettinen & Nurminen method; Test type: Superiority; p < 0.001, Miettinen & Nurminen — p-value is 1-sided; Percentage Point Difference = 85.2, 95% CI 2-sided [82.3 to 87.7] — V114-Prevnar 13™

15. Secondary Outcome: Anti-Pneumococcal Polysaccharide (Anti-PnP) Serotype-Specific Immunoglobulin G (IgG) Geometric Mean Concentrations (GMC) One Month After Vaccination 4 for 2 Unique V114 Seroptypes
Description: Serotype-specific anti-PnP GMCs were measured with PnECL. The GMC for each serotype is reported.
Time Frame: One month after Vaccination 4 (Month 13 to Month 16)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 858 | 856
ug/mL
  22F: number analyzed (Participants) | 714 | 682
  22F | 7.52 [7.09 to 7.98] | 0.11 [0.10 to 0.12]
  33F: number analyzed (Participants) | 714 | 677
  33F | 4.15 [3.89 to 4.42] | 0.09 [0.09 to 0.10]
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 68.80, 95% CI 2-sided [63.10 to 75.02] — V114/Prevnar 13™
Statistical Analysis 2: Comparison: V114 vs Prevnar 13™; [analysis description as in outcome 13, analysis 2]; Test type: Superiority; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 44.91, 95% CI 2-sided [41.04 to 49.14] — V114/Prevnar 13™

16. Secondary Outcome: Anti-Pneumococcal Polysaccharide (Anti-PnP) Serotype-Specific Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMT) One Month After Vaccination 3
Description: Serotype-specific anti-PnP OPA GMTs were measured with multiplex opsonophagocytic assay (MOPA). The GMTs for each serotype are summarized.
Time Frame: One month after Vaccination 3 (Month 7)
Population: Due to the large serum volume required for MOPA, the analysis population for OPA testing was performed on a subset of participants, which included the first 20% of all participants with sufficient serum volume at 30 days post-dose 3.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 176 | 168
Titers
  Serotype 1: number analyzed (Participants) | 170 | 162
  Serotype 1 | 56.9 [46.1 to 70.3] | 78.3 [61.5 to 99.5]
  Serotype 3: number analyzed (Participants) | 169 | 158
  Serotype 3 | 284.7 [253.5 to 319.8] | 210.6 [188.2 to 235.7]
  Serotype 4: number analyzed (Participants) | 169 | 159
  Serotype 4 | 1304.8 [1139.6 to 1494.0] | 1566.7 [1381.8 to 1776.4]
  Serotype 5: number analyzed (Participants) | 171 | 162
  Serotype 5 | 387.4 [315.0 to 476.3] | 510.8 [415.9 to 627.2]
  Serotype 6A: number analyzed (Participants) | 171 | 159
  Serotype 6A | 2072.1 [1787.5 to 2401.9] | 2743.4 [2368.1 to 3178.2]
  Serotype 6B: number analyzed (Participants) | 169 | 160
  Serotype 6B | 1932.5 [1612.1 to 2316.6] | 1963.7 [1604.9 to 2402.8]
  Serotype 7F: number analyzed (Participants) | 170 | 158
  Serotype 7F | 4973.2 [4277.6 to 5781.8] | 7335.1 [6181.8 to 8703.5]
  Serotype 9V: number analyzed (Participants) | 168 | 162
  Serotype 9V | 1217.3 [1040.2 to 1424.6] | 1534.1 [1305.5 to 1802.8]
  Serotype 14: number analyzed (Participants) | 167 | 160
  Serotype 14 | 2400.7 [1980.8 to 2909.6] | 1853.1 [1511.2 to 2272.5]
  Serotype 18C: number analyzed (Participants) | 171 | 162
  Serotype 18C | 1171.2 [1022.7 to 1341.4] | 1330.2 [1158.3 to 1527.5]
  Serotype 19A: number analyzed (Participants) | 171 | 162
  Serotype 19A | 841.3 [716.0 to 988.6] | 1400.7 [1205.5 to 1627.4]
  Serotype 19F: number analyzed (Participants) | 171 | 162
  Serotype 19F | 703.9 [614.2 to 806.6] | 850.6 [744.5 to 971.9]
  Serotype 23F: number analyzed (Participants) | 167 | 158
  Serotype 23F | 2078.9 [1779.2 to 2428.9] | 3668.8 [3069.2 to 4385.6]
  Serotype 22F: number analyzed (Participants) | 170 | 155
  Serotype 22F | 1849.3 [1606.9 to 2128.2] | 9.1 [7.9 to 10.4]
  Serotype 33F: number analyzed (Participants) | 170 | 155
  Serotype 33F | 8262.6 [6585.3 to 10367.1] | 119.6 [83.2 to 171.8]

17. Secondary Outcome: Anti-Pneumococcal Polysaccharide (Anti-PnP) Serotype-Specific Opsonophagocytic Activity (OPA) Response Rates One Month After Vaccination 3
Description: Serotype-specific anti-PnP OPA GMTs were measured with MOPA. The percentage of participants meeting ≥0.35 ug/mL are reported for each serotype.
Time Frame: One month after Vaccination 3 (Month 7)
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 176 | 168
Percentage of participants
  Serotype 1: number analyzed (Participants) | 170 | 162
  Serotype 1 | 86.5 [80.4 to 91.2] | 87.7 [81.6 to 92.3]
  Serotype 3: number analyzed (Participants) | 169 | 158
  Serotype 3 | 100.0 [97.8 to 100.00] | 100.0 [97.7 to 100.0]
  Serotype 4: number analyzed (Participants) | 169 | 159
  Serotype 4 | 99.4 [96.7 to 100.0] | 100.0 [97.7 to 100.0]
  Serotype 5: number analyzed (Participants) | 171 | 162
  Serotype 5 | 96.5 [92.5 to 98.7] | 98.1 [94.7 to 99.6]
  Serotype 6A: number analyzed (Participants) | 171 | 159
  Serotype 6A | 97.1 [93.3 to 99.0] | 98.1 [94.6 to 99.6]
  Serotype 6B: number analyzed (Participants) | 169 | 160
  Serotype 6B | 98.2 [94.9 to 99.6] | 98.1 [94.6 to 99.6]
  Serotype 7F: number analyzed (Participants) | 170 | 158
  Serotype 7F | 100.0 [97.9 to 100.0] | 100.0 [97.7 to 100.0]
  Serotype 9V: number analyzed (Participants) | 168 | 162
  Serotype 9V | 98.2 [94.9 to 99.6] | 97.5 [93.8 to 99.3]
  Serotype 14: number analyzed (Participants) | 167 | 160
  Serotype 14 | 98.8 [95.7 to 99.9] | 98.8 [95.6 to 99.8]
  Serotype 18C: number analyzed (Participants) | 171 | 162
  Serotype 18C | 98.8 [95.8 to 99.9] | 99.4 [96.6 to 100.00]
  Serotype 19A: number analyzed (Participants) | 171 | 162
  Serotype 19A | 98.2 [95.0 to 99.6] | 99.4 [96.6 to 100.0]
  Serotype 19F: number analyzed (Participants) | 171 | 162
  Serotype 19F | 95.9 [91.7 to 98.3] | 98.8 [95.6 to 99.9]
  Serotype 23F: number analyzed (Participants) | 167 | 158
  Serotype 23F | 99.4 [96.7 to 100.0] | 100.0 [97.7 to 100.0]
  Serotype 22F: number analyzed (Participants) | 170 | 155
  Serotype 22F | 99.4 [96.8 to 100.0] | 5.8 [2.7 to 10.7]
  Serotype 33F: number analyzed (Participants) | 170 | 155
  Serotype 33F | 98.8 [95.8 to 99.9] | 56.8 [48.6 to 64.7]

18. Secondary Outcome: Anti-Pneumococcal Polysaccharide (Anti-PnP) Serotype 3-Specific Immunoglobulin G (IgG) Response Rate One Month After Vaccination 3
Description: Serotype 3-specific anti-PnP IgG response rates were measured with PnECL. The percentage of participants with IgG Ab ≥0.35 ug/mL are reported for Serotype 3.
Time Frame: One month after Vaccination 3 (Month 7)
Population: All randomized participants who did not have protocol deviations that could have substantially affected the results of the immunogenicity analysis, who had sufficient blood volume to perform the analysis, and who had available serotype 3-specific IgG data.
Measure: Number; unit: Percentage of participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 699 | 662
Percentage of participants | 94.7 | 79.2
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Estimated difference, CI, and p-value are based on the Miettinen & Nurminen method; Test type: Superiority; p < 0.001, Miettinen & Nurminen — p-value is 1-sided; Percentage Point Difference = 15.6, 95% CI 2-sided [12.1 to 19.2] — V114-Prevnar 13™

19. Secondary Outcome: Anti-Pneumococcal Polysaccharide (Anti-PnP) Serotype 3-Specific Immunoglobulin G (IgG) Geometric Mean Concentration (GMC) One Month After Vaccination 3
Description: Serotype 3-specific anti-PnP GMC was measured with PnECL.
Time Frame: One month after Vaccination 3 (Month 7)
Population: as for outcome 18
Measure: Geometric Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 699 | 662
ug/mL | 1.08 [1.03 to 1.14] | 0.62 [0.59 to 0.66]
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; GMC ratio, CI, and p-value are calculated using the t-distribution with the variance estimate from a serotype-specific linear model utilizing the natural log-transformed antibody concentrations as the response and a single term for vaccination group; Test type: Superiority; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 1.73, 95% CI 2-sided [1.61 to 1.87] — V114/Prevnar 13™

20. Secondary Outcome: Anti-Pneumococcal Polysaccharide (Anti-PnP) Serotype 3-Specific Immunoglobulin G (IgG) Geometric Mean Concentration (GMC) One Month After Vaccination 4
Description: Serotype 3-specific anti-PnP GMC were measured with PnECL.
Time Frame: One month after Vaccination 4 (Month 13 to Month 16)
Population: All randomized participants who did not have protocol deviations that could have substantially affected the results of the immunogenicity analysis who had sufficient blood volume to perform the analysis, and who had available serotype 3-specific IgG data.
Measure: Geometric Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 712 | 686
ug/mL | 0.96 [0.91 to 1.01] | 0.71 [0.67 to 0.75]
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; [analysis description as in outcome 19, analysis 1]; Test type: Superiority; p < 0.001, t-test, 1 sided; GMC Ratio (V114 / Prevnar 13™) = 1.35, 95% CI 2-sided [1.25 to 1.46] — V114/Prevnar 13™

ADVERSE EVENTS:
Time Frame: Non-serious AEs (NSAEs): Up to ~14 days after each vaccination; SAEs and all-cause mortality: Up to ~6 months after Vaccination 4 (up to ~21 months)
Description: All-cause mortality was analyzed in all randomized participants; SAEs and NSAEs were analyzed in all randomized participants who received at least 1 dose of study vaccination with follow-up after V114 or Prevnar 13™.
Groups:
- Cross-treated Participants: One participant assigned to the Prevnar 13™ arm who inadvertently received both V114 and Prevnar 13™. The participant received a single 0.5 mL IM injection of Prevnar 13™ on Day 1 between 42-90 days of age inclusive (Vaccination 1), Month 4 from 4 months of age to 1 day prior to 5 months of age (Vaccination 2), Month 6 from 6 months of age to 1 day prior to 7 months of age (Vaccination 3) and a single 0.5 mL IM injection of V114 Months 12-15 from 12 months of age to 1 day prior to 16 months of age (Vaccination 4). The participant concomitantly received other licensed paediatric vaccines as follows: RotaTeq™, Pentacel™, RECOMBIVAX HB™ on Day 1, Month 4, and Month 6; VAQTA™, HIBERIX™, M-M-R™ II, VARIVAX™ on Months 12-15.
Arm/Group | V114 | Prevnar 13™ | Cross-treated Participants
All-Cause Mortality (participants affected / at risk) | 1/860 | 1/859 | 0/1
Serious Adverse Events (participants affected / at risk) | 88/858 | 81/855 | 1/1
Other Adverse Events (participants affected / at risk) | 790/858 | 778/855 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (N=858) | Prevnar 13™ (N=855) | Cross-treated Participants (N=1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Heart disease congenital (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 3 (3) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 11 (12) | 6 (6) | 1 (1)
Bronchitis (Infections and infestations) | 5 (5) | 2 (2) | 0 (0)
Bronchitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Croup infectious (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Enterovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Exanthema subitum (Infections and infestations) | 3 (3) | 3 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 7 (7) | 11 (13) | 0 (0)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 6 (6) | 2 (2) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpangina (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 5 (5) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 4 (4) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 7 (7) | 12 (12) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Scarlet fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 3 (3) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral diarrhoea (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 4 (4) | 2 (2) | 0 (0)
Viral rash (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Viral rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 3 (4) | 2 (2) | 0 (0)
Idiopathic generalised epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Infantile spasms (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Penile haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Kawasaki's disease (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (N=858) | Prevnar 13™ (N=855) | Cross-treated Participants (N=1)
Diarrhoea (Gastrointestinal disorders) | 46 (62) | 62 (76) | 0 (0)
Vomiting (Gastrointestinal disorders) | 42 (54) | 46 (52) | 0 (0)
Injection site erythema (General disorders) | 289 (488) | 329 (584) | 1 (1)
Injection site induration (General disorders) | 226 (385) | 229 (404) | 1 (1)
Injection site pain (General disorders) | 427 (903) | 401 (832) | 1 (2)
Injection site swelling (General disorders) | 226 (360) | 205 (348) | 0 (0)
Pyrexia (General disorders) | 265 (431) | 270 (464) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 55 (55) | 42 (44) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 294 (579) | 308 (606) | 0 (0)
Somnolence (Nervous system disorders) | 506 (1257) | 530 (1309) | 0 (0)
Irritability (Psychiatric disorders) | 656 (2514) | 645 (2435) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 35 (39) | 45 (48) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 36 (40) | 47 (49) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 56 (69) | 56 (69) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-16): https://cdn.clinicaltrials.gov/large-docs/48/NCT03893448/Prot_SAP_000.pdf